CLINICAL TRIAL: NCT06942676
Title: The Effects of Core Exercises on Change of Direction, Vertical Jump, Sprint, and Postural Sway: An Experimental Study
Brief Title: Core Exercises and Their Effects on Sprint, Jump, Agility, and Balance in Amateur Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORE2025-SK
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Athletic Performance Improvement Through Core Training
Keywords: Core Training; Sprint; Vertical jump; Postural sway; change of direction

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two arms: (1) Core training group, which performed a 4-week structured core exercise program in addition to their routine training; (2) Control group, which continued regular training without additional intervention.
Masking Description: Due to the nature of the exercise intervention, no blinding was applied. Both participants and investigators were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Training Group (Experimental): Participants in this group received a 4-week core training program in addition to their regular soccer training. The program included dynamic and static core stabilization exercises, performed 3 times per week, each session lasting approximately 25-30 minutes.
  Interventions: Behavioral: Core Exercise Program
- Control Group (No Intervention): Participants in this group continued their usual soccer training routine and did not receive any additional core training during the 4-week period.

INTERVENTIONS:
Behavioral: Core Exercise Program — This intervention consists of a 4-week core training program including exercises like planks, side planks, bird-dogs, bridges, and dead bugs, performed 3 days per week alongside regular soccer training. Each session lasted approximately 25-30 minutes.
  Arms: Core Training Group

SUMMARY:
This study aimed to investigate the effects of a 4-week core exercise program on sprint, vertical jump, agility, and postural sway performance in amateur male soccer players aged 18-23. Participants were randomly assigned to an intervention group (core training) or a control group (regular training). Physical performance tests were conducted before and after the training program. The results are expected to help coaches and sports scientists better understand the performance benefits of core training.

DETAILED DESCRIPTION:
This randomized controlled study investigated the effects of a 4-week core exercise program on sprint, vertical jump, agility, and postural sway performance in amateur male soccer players aged 18 to 23. Thirty participants were randomly assigned to either a core training group (n=15) or a control group (n=15). The core training group performed additional core stability exercises three times per week, while the control group continued their regular training routine. All participants completed physical performance tests, including 10- and 20-meter sprint, change of direction test, countermovement jump (CMJ), and postural sway assessment using a force platform. Pre- and post-test comparisons were conducted to evaluate the intervention's effectiveness. Ethical approval was obtained from the Gazi University Ethics Committee (Approval No: 2024-1685). The study was designed to help coaches and sport scientists understand how core training may improve athletic performance parameters in amateur football players.

ELIGIBILITY:
Inclusion Criteria:

* Male amateur soccer players aged 18 to 23 years
* Actively participating in regular soccer training (minimum 3 sessions/week)
* No musculoskeletal injuries within the last 6 months
* Provided informed consent

Exclusion Criteria:

* History of lower extremity surgery
* Any neurological or vestibular disorders
* Participation in core training within the past 3 months
* Use of medication that may affect balance or neuromuscular performance

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change of Direction Performance (Illinois Test) | Baseline (Week 0) and Week 5 (immediately after the 4-week intervention)
  Change of direction (COD) performance was measured using the Illinois Change of Direction Test. Participants completed the test before and after a 4-week core training intervention. COD time was recorded using infrared timing gates, and the best of two attempts was used for analysis. Lower completion time indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Selman Kaya, Phd, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there is no definitive plan for individual participant data (IPD) sharing. The decision will depend on future institutional policies, ethical approvals, and data availability.